CLINICAL TRIAL: NCT03336931
Title: A Multicenter Prospective Study of the Feasibility and Clinical Value of a Diagnostic Service for Identifying Therapeutic Targets and Recommending Personalised Treatment for Children and Adolescents With High-risk Cancer
Brief Title: PRecISion Medicine for Children With Cancer
Acronym: PRISM
Status: Active, not recruiting | Type: Observational
Sponsor: Sydney Children's Hospitals Network (Other)
Collaborators: Children's Cancer Institute Australia (Unknown); Australian & New Zealand Children's Haematology/Oncology Group (Other); Garvan Institute of Medical Research (Other); German Cancer Research Center (Other)
Responsible Party: Principal Investigator, Dr David Ziegler, Professor, Sydney Children's Hospitals Network
Other Study IDs: PRISM
Record Dates: First submitted 2017-10-22; First posted 2017-11-08 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Childhood Cancer; Childhood Solid Tumor; Childhood Brain Tumor; Childhood Leukemia; Refractory Cancer; Relapsed Cancer
Keywords: children; precision medicine; personalised medicine; high-risk cancer; refractory; recurrent; sequencing; patient derived xenograft; molecular profiling; paediatric
MeSH Terms: conditions — Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh, cryopreserved or frozen tumor, bone marrow or blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High-risk childhood cancers: Expected survival < 30%
  Interventions: Diagnostic Test: Molecular profiling and drug testing

INTERVENTIONS:
Diagnostic Test: Molecular profiling and drug testing — 1. Laboratory analysis including:
     A. Tumour molecular profiling: targeted whole exon variant analysis, whole genome (DNA) and transcriptome (RNA) sequencing, methylation analysis, proteomics analysis, immunohistochemistry B. In vitro high-throughput drug sensitivity testing C. In vivo drug testing using patient-derived xenograft (PDX) models D. Liquid biopsies
  2. Multi-disciplinary Tumour Board case discussion
  3. Recommendation of personalised therapy

SUMMARY:
This is a multicentre prospective study of the feasibility and clinical value of a diagnostic service for identifying therapeutic targets and recommending personalised treatment for children and adolescents with high-risk cancer.

DETAILED DESCRIPTION:
This is a multicentre study conducted under the Zero Childhood Cancer Program. The study will be enrolling patients under the age of 21 with high-risk cancer over 3 years from cancer centres in Australia. Patient's cancer cells will be tested for genetic abnormalities (mutations) and undergoing drug testing in highly specialised laboratories. A Multidisciplinary Tumour Board comprising of oncologists, clinical geneticists and scientists will then discuss the results of each case and determine whether a personalised medicine recommendation can be made. A report describing the results and Tumour Board recommendation (if any) will be provided to the patient's treating doctor. It is always at the discretion of the treating doctor whether to alter the patient's management based on the information arising from this research project.

ELIGIBILITY:
Inclusion criteria (all must be met)

1. Age ≤ 21 years
2. Histologic diagnosis of high-risk malignancy defined as expected overall survival < 30% OR where standard therapy would result in unacceptable and severe morbidity
3. Appropriate tissue samples are available for analysis
4. Life expectancy > 6 weeks
5. Written informed consent

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Paediatric patients who are being treated for high-risk cancer in Australia
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2017-09-05 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Personalized medicine recommendation | 5 years
  Proportion of patients for whom personalized medicine recommendation can be made using a comprehensive diagnostic platform within a clinically relevant timeframe

SECONDARY OUTCOMES:
Tumor samples with actionable molecular alterations | 5 years
  Proportion of tumor samples found to have actionable molecular alterations
Successfully conducted in vitro high throughput drug screening and in vivo drug sensitivity testing | 5 years
  Proportion of tumours where in vitro high throughput drug screening and in vivo drug sensitivity testing can be successfully performed
Identification of potential treatment by in vitro or in vivo drug screening | 5 years
  Proportion of tumors for which a potential treatment option is identified by in vitro or in vivo drug screening
Reporting turnaround time | 5 years
  Number of weeks from enrollment to issuing a report to the treating clinician
Patients receiving the recommended personalized therapy | 5 years
  Proportion of patients who subsequently receive the recommended personalized therapy
Barriers or reasons for patients not receiving the recommended personalized therapy | 5 years
  Description of the barriers or reasons for patients not receiving the recommended personalized therapy

OTHER OUTCOMES:
Impact of personalized therapy on progression-free survival | Up to 5 years
  Time interval from enrollment until disease progression or death for patients who have received personalized therapy versus those who have not
Impact of personalized therapy on overall survival | Up to 5 years
  Time interval from enrollment until death for patients who have received personalized therapy versus those who have not

CONTACTS AND LOCATIONS:
Overall Officials: A/Prof David Ziegler, MBBS, Principal Investigator — Sydney Children's Hospitals Network
Locations (8):
- Australia (8):
  - John Hunter Children's Hospital, Newcastle, New South Wales
  - Sydney Children's Hospital, Randwick, Sydney, New South Wales
  - The Children's Hospital at Westmead, Sydney, New South Wales
  - Queensland Children's Hospital, Brisbane, Queensland
  - Women's and Children's Hospital, Adelaide, South Australia
  - Royal Children's Hospital, Melbourne, Victoria
  - Monash Children's Hospital, Melbourne, Victoria
  - Perth Children's Hospital, Perth, Western Australia

REFERENCES:
- [Derived] Robertson EG, Hetherington K, Hunter JD, McGillycuddy M, Venkatesha V, Lau LMS, Khuong-Quang DA, Ziegler DS, Wakefield CE. Whatever It Takes: Parents' Perspectives of Patient-Derived Xenograft Mouse Models for Poor Prognosis Childhood Cancer. JCO Precis Oncol. 2025 Apr;9:e2400840. doi: 10.1200/PO-24-00840. Epub 2025 Apr 10. PMID 40209140
- [Derived] Lau LMS, Khuong-Quang DA, Mayoh C, Wong M, Barahona P, Ajuyah P, Senapati A, Nagabushan S, Sherstyuk A, Altekoester AK, Fuentes-Bolanos NA, Yeung V, Sullivan A, Omer N, Diamond Y, Jessop S, Battaglia L, Zhukova N, Cui L, Lin A, Gifford AJ, Fleuren EDG, Dalla-Pozza L, Moore AS, Khaw SL, Eisenstat DD, Gottardo NG, Wood PJ, Tapp H, Alvaro F, McCowage G, Nicholls W, Hansford JR, Manoharan N, Kotecha RS, Mateos MK, Lock RB, Tyrrell V, Haber M, Trahair TN, Cowley MJ, Ekert PG, Marshall GM, Ziegler DS. Precision-guided treatment in high-risk pediatric cancers. Nat Med. 2024 Jul;30(7):1913-1922. doi: 10.1038/s41591-024-03044-0. Epub 2024 Jun 6. PMID 38844796
- [Derived] Ajuyah P, Mayoh C, Lau LMS, Barahona P, Wong M, Chambers H, Valdes-Mora F, Senapati A, Gifford AJ, D'Arcy C, Hansford JR, Manoharan N, Nicholls W, Williams MM, Wood PJ, Cowley MJ, Tyrrell V, Haber M, Ekert PG, Ziegler DS, Khuong-Quang DA. Histone H3-wild type diffuse midline gliomas with H3K27me3 loss are a distinct entity with exclusive EGFR or ACVR1 mutation and differential methylation of homeobox genes. Sci Rep. 2023 Mar 7;13(1):3775. doi: 10.1038/s41598-023-30395-4. PMID 36882456
- [Derived] Rapport F, Smith J, O'Brien TA, Tyrrell VJ, Mould EV, Long JC, Gul H, Braithwaite J. Development of an implementation and evaluation strategy for the Australian 'Zero Childhood Cancer' (Zero) Program: a study protocol. BMJ Open. 2020 Jun 23;10(6):e034522. doi: 10.1136/bmjopen-2019-034522. PMID 32580982